CLINICAL TRIAL: NCT07228832
Title: A Randomized, Active-Controlled, Double-blind, Multicenter, Phase 3 Clinical Study of Ivonescimab in Combination With FOLFOX Versus Bevacizumab in Combination With FOLFOX for the First-line Treatment of Metastatic Colorectal Cancer
Brief Title: Phase III Study of Ivonescimab or Bevacizumab Combined With FOLFOX in Patients With Metastatic Colorectal Cancer
Acronym: HARMONi-GI3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMT112-3005
Record Dates: First submitted 2025-11-10; First posted 2025-11-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer (CRC)
Keywords: mCRC; Ivonescimab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Ivonescimab in combination with mFOLFOX6 (Experimental): Subjects will receive Ivonescimab Plus mFOLFOX6 via intravenous infusion (IV) Q2W, up to 8 cycles. Afterward, Ivonescimab plus Leucovorin and 5-FU will be used for maintenance treatment (administered on Day 1 of each cycle, Q2W) up to 2 years.
  Interventions: Drug: Drug: Ivonescimab Injection
- Arm B: Bevacizumab in combination with mFOLFOX6 (Active Comparator): Subjects will receive bevacizumab Plus mFOLFOX6 (Oxaliplatin, Leucovorin and 5-Fluorouracil) via intravenous infusion (IV) Q2W, up to 8 cycles in treatment periods per the randomization schedule. Afterward, bevacizumab Plus 5-FU and Leucovorin will be used for maintenance treatment (administered on Day 1 of each cycle, Q2W) up to 2 years.
  Interventions: Drug: Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: Drug: Ivonescimab Injection — Subjects will receive Ivonescimab Plus mFOLFOX6 (Oxaliplatin, Leucovorin and 5-Fluorouracil) via intravenous infusion (IV) Q2W, up to 8 cycles. Afterward, Ivonescimab plus Leucovorin and 5-Fluorouracil will be used for maintenance treatment (administered on Day 1 of each cycle, Q2W) for up to 2 years.
  Other Names: Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: Arm A: Ivonescimab in combination with mFOLFOX6
Drug: Drug: Bevacizumab Injection — Subjects will receive bevacizumab Plus mFOLFOX6 (Oxaliplatin, Leucovorin and 5-Fluorouracil) via intravenous infusion (IV) Q2W, up to 8 cycles in treatment periods per the randomization schedule. Afterward, bevacizumab Plus 5-FU and Leucovorin will be used for maintenance treatment (administered on Day 1 of each cycle, Q2W) up to 2 years.
  Other Names: Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: Arm B: Bevacizumab in combination with mFOLFOX6

SUMMARY:
A Randomized, Active-Controlled, Double-blind, Multicenter, Phase 3 Clinical Study of Ivonescimab in Combination with mFOLFOX6 (Oxaliplatin, Leucovorin and 5-Fluorouracil) versus Bevacizumab in Combination with FOLFOX for the First-line Treatment of Metastatic Colorectal Cancer(HARMONi-GI3)

DETAILED DESCRIPTION:
This trial will be performed as a phase 3, randomized, active-controlled, double-blind, multiregional study comparing Ivonescimab in combination with mFOLFOX6 (Oxaliplatin, Leucovorin and 5-Fluorouracil) versus Bevacizumab in combination with mFOLFOX6 in patients with metastatic colorectal cancer who have not previously received systemic therapy for metastatic disease. Approximately 600 patients will be randomly assigned to the 2 treatment groups in a 1:1 ratio. Each enrolled subject will receive an intravenous infusion of the Ivonescimab/Bevacizumab Plus mFOLFOX6 (Q2W, up to 8 cycles) in treatment periods per the randomization schedule. Afterward, Ivonescimab/ Bevacizumab Plus 5-Fluorouracil and Leucovorin will be used for maintenance treatment (administered on Day 1 of each cycle, Q2W) for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status score of 0 or 1
2. Expected life expectancy ≥ 6 months
3. Patients with histologically or cytologically confirmed metastatic CRC
4. No prior systemic therapy for metastatic CRC
5. At least 1 measurable noncerebral lesion

Exclusion Criteria:

1. Microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) disease
2. Known BRAF V600E mutant status
3. Current presence of significant radiographic or clinical manifestations of gastrointestinal (GI) obstruction
4. Ascites requiring paracentesis within last 30 days
5. Patients who have received prior immunotherapy or anti-angiogenic therapy for colorectal cancer
6. Active or prior history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
7. Resectable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
PFS by IRRC based on RECIST v1.1 | Up to approximately 2.5 years
  Progression-free survival (PFS) assessed by IRRC per RECIST v1.1

SECONDARY OUTCOMES:
Overall Survival (OS) in the population | Up to approximately 4 years
  Overall Survival (OS) in the mCRC population
ORR | Up to approximately 2.5 years
  Efficacy measures such as overall response rate (ORR), which is the proportion of subjects with CR or PR by IRRC based on RECIST v1.1
Adverse Events (AE) | Up to approximately 4 years
  incidence and severity of adverse events (AEs) and clinically significant abnormal laboratory test results [From the time subject signs the ICF to 30 days (AE) and 90 days (SAE related to ivonescimab/bevacizumab) after the last dose of study treatment or initiation of other anticancer therapy, whichever occurs first]
DoR | up to approximately 2.5 years
  Efficacy measures such as duration of response (DoR), which is the proportion of subjects with CR or PR by IRRC based on RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Clinical Study Site, Cerritos, California
  - Clinical Study Site, Los Angeles, California
  - Clinical Study Site, Murrieta, California
  - Clinical Study Site, Hialeah, Florida
  - Clinical Study Site, Port Saint Lucie, Florida
  - Clinical Study Site, O'Fallon, Illinois
  - Clinical Study Site, Saint Louis Park, Minnesota
  - Clinical Study Site, Lincoln, Nebraska
  - Clinical Study Site, Spokane, Washington